CLINICAL TRIAL: NCT01931280
Title: A Transgenerational e-Intervention for Gestational Diabetics and Their Offspring: A Pilot Trial
Brief Title: A Transgenerational e-Intervention for Gestational Diabetics and Their Offspring
Acronym: GooD MomS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-0827; 1R21DK095189-01 (NIH)
Record Dates: First submitted 2013-08-22; First posted 2013-08-29 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2014-09

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy
Keywords: Gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Counseling (Experimental): Participants will obtain access to an internet-based educational intervention.
  Interventions: Behavioral: Lifestyle Counseling
- Usual Care (Self-Directed) (No Intervention): Participants receive information via email on health related topics that surround pregnancy, physical activity, nutrition, and gestational diabetes.

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Participants receive lifestyle counseling on healthy eating and physical activity through an internet based program or self-directed educational program.
  Other Names: Healthy Lifestyle; Glucose Control
  Arms: Lifestyle Counseling

SUMMARY:
This study includes a behavioral educational intervention that focuses on healthy eating, physical activity and glucose management during pregnancy and post partum among women newly diagnosed with gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
This is a pilot trial in which 50 women newly diagnosed with gestational diabetes are randomized to either one of two groups: 1) active internet intervention or 2)Usual Care (Self-directed) educational intervention. The primary pregnancy outcome is change in A1C. The primary postpartum outcome is weight.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gestational diabetes Confirmed singleton pregnancy 24-32 weeks gestation age Planning to deliver within the study area

Exclusion Criteria:

* Pre-existing diabetes (type 1 or 2) Non-english speaking Not planning to deliver in the study area

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin | Baseline and 36 weeks gestation

SECONDARY OUTCOMES:
Change in weight after pregnancy | 6 weeks postpartum to 30 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Wanda K. Nicholson, MD MPH MBA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Setse R, Grogan R, Cooper LA, Strobino D, Powe NR, Nicholson W. Weight loss programs for urban-based, postpartum African-American women: perceived barriers and preferred components. Matern Child Health J. 2008 Jan;12(1):119-27. doi: 10.1007/s10995-007-0211-6. Epub 2007 Jun 7. PMID 17554614